CLINICAL TRIAL: NCT06150443
Title: Pilot Study Evaluating the Elasticity and Shear Wave Modulus (Stiffness) of the Median Nerve in Patients With Mild to Moderate Idiopathic Carpal Tunnel Syndrome Receiving OMT and Conservative Therapy
Acronym: COMET-AOA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kettering Health Network (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHN-2023-130
Record Dates: First submitted 2023-11-14; First posted 2023-11-29 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Manipulation, Osteopathic; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - OMT Only (Experimental): Osteopathic manipulative treatment will include the interosseous membrane technique, the flexor retinaculum soft tissue technique, and the radiocarpal somatic dysfunction technique. The cervical spine will also be treated, with particular attention to the C5-7 levels, all the way to the wrist and hand as the physician sees fit based on the findings of the osteopathic structural exam.
  Interventions: Other: Osteopathic manipulative treatment (OMT)
- Group 2 - OMT + Conservative Treatment (Active Comparator): Will receive Osteopathic manipulative treatment in addition to conservative treatment. Conservative therapy will be defined as including the use of splints, NSAIDs, opioids, and therapeutic injection of the carpal tunnel with steroids. Physical and Occupational therapy will be excluded from the conservative therapy regimen. Osteopathic manipulative treatment will include the interosseous membrane technique, the flexor retinaculum soft tissue technique, and the radiocarpal somatic dysfunction technique. The cervical spine will also be treated, with particular attention to the C5-7 levels, all the way to the wrist and hand as the physician sees fit based on the findings of the osteopathic structural exam.
  Interventions: Other: Osteopathic manipulative treatment (OMT); Other: Conservative treatment
- Group 3 - Conservative Treatment Only (Active Comparator): Conservative therapy will be defined as including the use of splints, NSAIDs, opioids, and therapeutic injection of the carpal tunnel with steroids. Physical and Occupational therapy will be excluded from the conservative therapy regimen.
  Interventions: Other: Conservative treatment

INTERVENTIONS:
Other: Osteopathic manipulative treatment (OMT) — Two osteopathic primary care physicians will performing osteopathic manipulative techniques with a minimum of three direct techniques focused on carpal tunnel. These techniques will include the interosseous membrane technique, the flexor retinaculum soft tissue technique, and the radiocarpal somatic dysfunction technique. They will also evaluate and treat the cervical spine, with particular attention to the C5-7 levels, all the way to the wrist and hand as they see fit based on the findings of their osteopathic structural exam.
  Arms: Group 1 - OMT Only; Group 2 - OMT + Conservative Treatment
Other: Conservative treatment — Conservative therapy will be defined as including the use of splints, NSAIDs, opioids, and therapeutic injection of the carpal tunnel with steroids. Physical therapy will be excluded from the conservative therapy regimen.
  Arms: Group 2 - OMT + Conservative Treatment; Group 3 - Conservative Treatment Only

SUMMARY:
To evaluate and quantify changes in the elasticity and shear wave modulus (stiffness) of the median nerve in patients diagnosed with mild to moderate carpal tunnel syndrome following osteopathic manipulative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral or bilateral mild to moderate carpal tunnel syndrome, based on recent EMG findings

Exclusion Criteria:

* History of undergoing recent physical therapy for treatment of carpal tunnel syndrome
* History of wrist trauma or surgery
* Hypothyroidism
* Severe CTS that has progressed to muscle atrophy
* Systemic disease or condition including but not limited to diabetes mellitus, thyroid disorders, rheumatoid disorders, Paget's bone disease, gout, myxedema, multiple myeloma, acromegaly, hepatic disease, dialysis patients, or other diseases or conditions in which peripheral neuropathies are common.
* Secondary cause of CTS such as a ganglion cyst, mass, or an accessory muscle shown by US or MRI of the affected wrist.
* Bifid median nerve as shown by US or MRI of the affected wrist
* pregnant or recently postpartum

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Elasticity of median nerve at the carpal tunnel inlet | baseline, post 2-week treatment, post 4-week treatment, post 6-week treatment
  Measured by shear wave elastography.
Cross-sectional area of median nerve in 3 locations | baseline, post 2-week treatment, post 4-week treatment, post 6-week treatment
  Measured by real-time grayscale ultrasound
Quick DASH Patient Survey Score | Completed at treatment visits (initial, 2 weeks, 4 weeks, and 6 weeks)
  This questionnaire asks the patient about their symptoms as well as their ability to perform certain activities. The QuickDASH, published in 2005 in the Journal of Bone and Joint Surgery, is a subset of 11 items from the 30-item DASH and is a self-reported questionnaire in which the response options are presented as 5-point Likert scales. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb.
CTS-6 Evaluation Tool Score | Completed at treatment visits (initial, 2 weeks, 4 weeks, and 6 weeks)
  The Value Added by Electrodiagnostic Testing in the Diagnosis of Carpal Tunnel Syndrome completed by the clinician. A score >12 = 0.80 probability of Carpal Tunnel Syndrome and a score >5 = 0.25 probability of Carpal Tunnel Syndrome.
Elasticity of the transverse carpal ligament | baseline, post 2-week treatment, post 4-week treatment, post 6-week treatment
  Measured by shear wave elastography.
Elasticity of the subsynovial connective tissue in the carpal tunnel | baseline, post 2-week treatment, post 4-week treatment, post 6-week treatment
  Measured by shear wave elastography.

SECONDARY OUTCOMES:
Motor Distal Latency | Baseline and at 8 weeks (end of study)
  Time it takes for an impulse to traverse the segment nearest the muscle.
Sensory Distal Latency | Baseline and at 8 weeks (end of study)
  Time it takes for an impulse to traverse the segment nearest the muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Gazaille, DO, Principal Investigator — Kettering Health
Locations (1):
- Kettering Health, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No